CLINICAL TRIAL: NCT02290964
Title: Effect of Acute Normovolemic Haemodilution on Allogenic Transfusion Needs in Patients Undergoing Laparotomy Surgery
Brief Title: Effect of Acute Normovolemic Haemodilution on Allogenic Transfusion Needs In Laparotomy
Acronym: ANH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitas Padjadjaran (Other)
Responsible Party: Principal Investigator, Tatang Bisri, Professor in anesthesiology, MD., PhD, Universitas Padjadjaran
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AN-201409.01
Record Dates: First submitted 2014-09-28; First posted 2014-11-14 (Estimated); Last update posted 2014-11-14 (Estimated); Status verified 2014-11

CONDITIONS: Surgery
Keywords: Acute normovolemic hemodilution; allogeneic transfusion

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control group (No Intervention): After general anesthesia is applied, surgery is performed. Whenever transfusion is indicated, the patients will received allogenic blood transfusion
- ANH group (Active Comparator): After general anesthesia is applied, blood from patients in this group were withdrawn. the volume of blood withdrawn was determined based on Gross equation. The blood obtained was then stored in the operating room at temperature between 23 - 25 Celsius degree, and given back to the patient whenever transfusion is indicated.
  Interventions: Procedure: ANH

INTERVENTIONS:
Procedure: ANH — After general anesthesia is applied, blood was taken through the cubital vein and collected into standard blood bags containing CPDA anti-coagulant. The blood obtained is then stored at temperature of 23 - 25 Celsius degree and given back to patients in the operating room after the bleeding stopped and as soon as there are indications of transfusion.
  Arms: ANH group

SUMMARY:
This study is aimed to determine if acute normovolemic hemodilution (ANH), an established blood conservation technique, reduces the requirement for allogeneic blood transfusion in operations with prediction of surgical bleeding over 20% of estimated blood volume (EBV)

DETAILED DESCRIPTION:
Allogeneic blood transfusion is often done during surgery to save life- threatening conditions. Blood conservation is a method that can reduce peri-operative allogeneic blood transfusion. This study has been conducted on 34 patients underwent laparotomy surgery with bleeding more than 20% of EBV. After being informed concent, research subjects were randomized into two groups: ANH (conducted ANH) and control group (without ANH). After starting general anesthesia, the ANH group was withdrawing blood based on Gross formula. Restoration of circulated volume was instituted by infusion of colloids. In control group, the operation was started right after the induction of anesthesia. The monitoring of blood pressure, heart rate, the amount of bleeding, total fluid, urine production, hemoglobin concentration and number of allogenic transfusion were recorded.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients scheduled for laparotomy under general anesthesia with potentially surgical bleeding > 20% of EBV
* ASA physical status I - II
* hemoglobin level before surgery > 11 g / dl for men and > 10 g / dl for women

Exclusion Criteria:

* impaired coagulation (INR> 1.5 and / or platelet count <100,000)
* active infection
* disruption of metabolic liver
* received anti fibrinolytic drugs

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2010-03; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Reduction of allogenic transfusion requirements | During surgery and 24 hours post surgery with target Hb > 8gr/dl
  The investigators evaluate number of patients require allogenic transfusion during surgery until 24 hours post surgery with targeted haemoglobin level > 8gr/dl. Blood pressure, heart rate, total bleeding, total fluid administration and urine production are also recorded in order to confirm that acute normovolemic haemodilution is safe in patients undergoing laparotomy surgery

CONTACTS AND LOCATIONS:
Overall Officials: Heni H Listianto, MD, Study Chair — Department of Anesthesiology and Therapy Intensive Faculty of Medicine Universitas Padjadjaran Dr. Hasan Sadikin General Hospital Bandung
Locations (1):
- Department of Anesthesiology and Therapy Intensive Faculty of Medicine/Dr. Hasan Sadikin General Hospital, Bandung, West Java, Indonesia